CLINICAL TRIAL: NCT02958540
Title: Randomized, Doubleblind, Placebo-controlled Trial in Healthy Adults of Safety and Immunogenicity of 2 Intranasal Doses of SynGEM®, an RSV Candidate Vaccine Containing F Glycoprotein Linked to a Bacterium-like-Particle (BLP) Carrier
Brief Title: Phase I Study for SynGEM, an Intranasal Respiratory Syncytial Virus (RSV) Prefusion F Subunit Candidate Vaccine
Acronym: SynGEM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mucosis BV (Industry)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MUC-SynGEM-001; 2015-003814-25 (EudraCT Number)
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Respiratory Syncytial Viral Infections
Keywords: Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SynGEM low dose (Experimental): Group 1: 18 subjects receiving SynGEM low dose
  Interventions: Biological: SynGEM
- SynGEM high dose (Experimental): Group 2: 18 subjects receiving SynGEM high dose
  Interventions: Biological: SynGEM
- placebo (Placebo Comparator): 12 subjects receiving placebo
  Interventions: Other: placebo

INTERVENTIONS:
Biological: SynGEM — Prime / boost vaccination in each group
  Arms: SynGEM high dose; SynGEM low dose
Other: placebo — prime /boost vaccination
  Arms: placebo

SUMMARY:
The study is a double-blind (within dose level), placebo-controlled Phase I study to assess the safety, reactogenicity and tolerability of two intranasal dose levels of SynGEM®: a low dose level (140 μg F-protein/2mg BLPs) and a high dose level ( 350 μg F-protein/5mg BLPs), each administered twice according to a prime-boost schedule 28 days apart at Day 1 and Day 29. The two dose levels will be recruited sequentially.

Immunogenicity end-points will include assessment of humoral and cellular responses at selected time-points.

DETAILED DESCRIPTION:
A total of 48 healthy adult volunteers aged 18 to 49 years will be recruited. The first 24 subjects will be randomized 3:1 to SynGEM® low dose level (140 μg F-protein/2mg BLPs) or placebo administered at Day 1 and Day 29 (Group 1). After completion of recruitment of Group 1, if no pausing rule is met until 7 days post prime in all Group 1 subjects, 24 additional subjects will be randomized 3:1 to SynGEM® high dose level (350 μg F-protein/2mg BLPs) or placebo administered at Day 1 and Day 29 (Group 2).

Recruitment will be guided by pre-specified pausing rules. Recruitment of Group 1 will be staggered as follows: a sentinel cohort of 2 subjects (1 subject receiving SynGEM® and 1 subject receiving placebo) will be recruited on study Day 1; subjects will be followed up to Visit 2 (3 days post-dosing) and if no pausing rule is met, a second cohort of 2 subjects (1 subject receiving SynGEM® and 1 subject receiving placebo) will be vaccinated; subjects will be followed up to Visit 2 (3 days post-dosing) and if no pausing rule is met, recruitment will be extended to the remaining 20 subjects (16 on SynGEM®/4 on placebo) of Group 1.

Escalation to the high dose level will be implemented only after collection of safety data of all subjects in Group 1 for at least 7 days post-prime if no pausing rule is met. Group 2 will also be comprised of a total of 24 subjects and recruitment will be staggered and subjected to the same pausing rules as in Group 1.

Each subject will return to the site for study visits 3, 7 and 28 days post-prime vaccination; 28 days after prime vaccination the boost vaccination will be administered and subjects will return 3, 7, 28 days after boost vaccination. A primary analysis will be carrying out on data collected up to this timepoints. Subjects will be followed up for safety and immunogenicity thereafter up to 180 days post-prime.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 - 49 years inclusive.
2. Able to give written informed consent to participate.
3. Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
4. Healthy, as determined by medical history, physical examination, vital signs, and clinical judgment.
5. Must have acceptable laboratory parameters* within 28 days before Day 1. Acceptable laboratory parameters are defined as follows:

   A. Hemoglobin, Red Blood Cell (RBC) count and hematocrit: within laboratory normal sex-specific range.

   B. White Blood Cell (WBC) count within the normal laboratory range C. Sodium and potassium within laboratory normal range D. Total bilirubin within laboratory normal range E. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST): ≤1.1x institutional ULN.

   F. Serum creatinine: ≤1.1x institutional upper limit of normal (ULN).

   *Note: If the acceptable laboratory screening parameters listed above are out of the above defined range, repeat of screening tests is permitted once, provided there is an alternative explanation for the out-of-range value. Out of range results for laboratory tests either listed or not in Section 8.6.3 other than those covered in the list above are acceptable if considered not clinically significant by the Investigator.
6. A Body Mass Index (BMI) between 18 and 32, inclusive. BMI = weight (kg)/height2 (m2).
7. Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and a negative urine β-hCG pregnancy test within 24 hours preceding receipt of each dose and agree to practice, if not already practicing, highly effective birth control measures from 28 days before the prime vaccination until at least 90 days after the boost vaccination. For women already practicing highly effective birth control measurements for at least 28 days at screening start, recruitment can occur as soon as all screening procedures are completed. The following birth control measure will be considered highly effective:

   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone releasing system, bilateral tubal ligation, vasectomized partner (if the partner is the sole sexual partner and has received medical assessment of the surgical success).
   2. True abstinence: when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception].
   3. If not heterosexually active at screening, must agree to practice highly effective birth control measures described above if they become heterosexually active from that moment onwards until at least 90 days after the boost vaccination.
   4. Agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction from the start of screening onwards until at least 90 days after the boost vaccination.
8. Women of non-childbearing potential, defined as postmenopausal (>45 years of age with amenorrhea for ≥2 years; for female of >45 years of age with amenorrhea for more than 6 months but less than 2 years confirmation of a serum follicle stimulating hormone (FSH) >40 mIU/mL will be required to consider them of non-childbearing potential) or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), are not required to use the birth control methods as described in Inclusion Criterion #7.
9. A man who has not had a vasectomy with medical assessment of the surgical success and is sexually active with a woman of childbearing potential must agree to consistently use a barrier method of birth control, such as condom with spermicidal foam/gel/film/cream/suppository. Men must also agree not to donate sperm from the first study vaccine administration (Day 1) until 90 days after the boost vaccination.
10. Subjects must be willing to provide verifiable identification and their National Insurance/Passport number for the purpose of The Over-volunteering Prevention System (TOPS) registration.
11. Subject must have a means to be contacted.

Exclusion Criteria:

1. History of acute respiratory disease in the 30 days preceding start of screening or documented infection with RSV in the previous 3 months.
2. Any chronic disease of the nasal cavity such as chronic hypertrophic or atrophic rhinitis, chronic sinusitis, ozena, Wegener's granulomatosis or granulomatosis with polyangiitis.
3. History of asthma or chronic obstructive pulmonary disease.
4. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic). This includes institution of a new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening.
5. Subjects who are positive for hepatitis B surface antigen, hepatitis C antibodies or HIV.
6. Pregnant or breastfeeding women, or planning to become pregnant while enrolled in the study or within 90 days after the boost vaccination.
7. Cancer, or treatment for cancer, within 3 years, excluding basal cell carcinoma or squamous cell carcinoma of the skin, which is allowed.
8. Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus.
9. Presently receiving or history of receiving, during the preceding 3-month period, any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulins, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable). Topical corticosteroids are allowed.
10. Receipt of any intranasal administration of drug or vaccine within the 30 days prior to the first administration of study vaccine or plans to receive any intranasal administration of drug or vaccine until the end of study visit.
11. Receipt of live attenuated vaccine within 30 days of first SynGEM® administration or plans to receive within 30 days after the last study vaccine administration, and receipt of any other vaccine within 15 days of first SynGEM® administration or plans to receive within 15 days after the last study vaccine administration.
12. Positive history of illicit drug use, of drug or alcohol abuse within the previous 6 months.
13. History of anaphylactic type reaction to injected vaccines.
14. History of allergic rhinitis or of allergy to food.
15. History of allergy to insect bites, latex, pollens, house dust mites that are considered significant by the Investigator.
16. Treatment with another investigational medicinal product (IMP) within 3 months prior to screening or with more than 2 IMPs in the past year.
17. Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the study period.
18. Loss of ˃ 500 mL blood within 3 months prior to screening.
19. Any major neurological disease, including migraine
20. Any condition that, in the Investigator's opinion, might interfere with the primary study objectives.
21. Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical examination) with or without fever, or a fever >38ºC does not represent an absolute exclusion criterion, but an exclusion criterion at that moment in time. Prime vaccination can be re-scheduled as deemed necessary by the Investigator.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessed through diaries for local and systemic tolerability and with follow up for occurrence of any adverse event | 7 days post each dose / 57 days post prime
  subjects' diary

SECONDARY OUTCOMES:
Immunogenicity responses | up to 180 day
  At baseline (day 1), Day 8, 29, 36, 57, 120, 180

CONTACTS AND LOCATIONS:
Overall Officials: Chris Chiu, PhD, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Centre for Translational and Experimental Medicine Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ascough S, Vlachantoni I, Kalyan M, Haijema BJ, Wallin-Weber S, Dijkstra-Tiekstra M, Ahmed MS, van Roosmalen M, Grimaldi R, Zhang Q, Leenhouts K, Openshaw PJ, Chiu C. Local and Systemic Immunity against Respiratory Syncytial Virus Induced by a Novel Intranasal Vaccine. A Randomized, Double-Blind, Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2019 Aug 15;200(4):481-492. doi: 10.1164/rccm.201810-1921OC. PMID 30753101